CLINICAL TRIAL: NCT01174758
Title: Development of an Instrumented System to Measure Mobility in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Fay B. Horak, Professor of Neurology, Oregon Health and Science University
Other Study IDs: 5029
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Parkinson's Disease
Keywords: balance; mobility; ON/OFF Levodopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Parkinson's disease: Individuals participating in the study have been diagnosed with idiopathic Parkinson's disease.

SUMMARY:
Developing technology to increase efficiency and decrease cost of clinical trials. The longterm objective of this project is to use new technologies to sensitively measure, automatically analyze and efficiently manage clinical trial data for Parkinson's disease (PD) and other neurological disorders. This project will focus on developing objective measures of balance and gait because mobility disability and falls are so critical for quality of life in PD. Clinical movement disorders experts will team up with a local start-up business to develop, produce, and test a novel clinical balance and gait assessment tool, the instrumented Timed Up and Go Test (iTUG) for patients with Parkinson's disease. Balance and gait will be measured with wireless sensors worn on the wrists, ankles and trunk while patients stand up from a chair, walk, turn and return to sit on the chair. Accelerations and angular velocities from the sensors will be automatically transmitted, stored, analyzed, and displayed as Mobility Scores on a remote, centralized computer, along with other patient information important for clinical trials. Specifically, this proposal will 1) create a commercially-available, clinical trial system that includes completely wireless sensor technology, a custom-made, user-friendly, computer interface and efficient data management server; 2) develop a mobility score from many potential balance and gait measures and 3) compare the sensitivity of the iTUG compared to traditional clinical tests of balance to changes in PD due to antiparkinson medication. By providing a more sensitive, accurate, and comprehensive method to quickly test and analyze balance and gait, clinical trials to improve mobility in patients with Parkinson's disease and other neurological disorders will be significantly more effective and efficient. This will permit clinical trials in Parkinson's disease to be completed with fewer subjects, shorter duration, and less cost.The current project will accelerate the development of new therapies for Parkinson's disease.

DETAILED DESCRIPTION:
The specific aims of the study:

Aim I. To create a novel, commercially-available system for mobility assessment in clinical trials for Parkinson's disease. We have already developed a laboratory prototype system for the iTUG test, but the computer interface, sensors, and data management system are too cumbersome for use in clinical trials. In this proposal, we will create a robust, user-friendly clinical system for the iTUG test using wireless inertial sensors and a new user interface developed by a Portland start-up company, Automated Parkinson's Disease Monitoring (APDM), headed by a co-investigator. This mobility measuring system will be integrated with a new centralized data management server also developed by APDM, Inc. to support automatic data analysis and data organization for multi-site clinical trials. The feasibility of the new, clinical system will then be vetted by using it in a busy Movement Disorders Clinic.

Aim II. To develop an objective, composite iTUG mobility score. We recently demonstrated that iTUG metrics are more sensitive in distinguishing mobility performance between people just diagnosed with PD from age-matched controls than traditional clinical tests. In this proposal, we will develop a composite mobility score from the iTUG gait and postural parameters most responsive to severity of PD and to the change from the levodopa ON and OFF states. The composite score will be calculated using statistical models that optimize differences in performance between 75 subjects with PD in the ON and OFF levodopa state.

Aim III. To prospectively determine the reliability, validity and responsiveness of the iTUG mobility score. We will perform a prospective study with 60 patients with PD that compares standard clinical measures of postural instability and gait difficulty mobility (PIGD items from the Unified Parkinson's Disease Rating Scale (UPDRS) and TUG stop-watch scores) with our new iTUG mobility score in the OFF and ON levodopa states. We hypothesize that the iTUG will have good test-retest reliability, be significantly correlated with standard clinical measures and fall history and be more responsive to dopaminergic state than current mobility tests used in clinical trials. This project will develop, produce, and test a novel clinical balance and gait assessment tool, the instrumented Timed Up and Go test (iTUG) using our new, wearable, inertial sensors and our new clinical trial data management server that automatically transmits, stores, and analyzes data collected with the iTUG. By automatically providing a more sensitive, accurate, and comprehensive method to test balance and gait, clinical trials to improve mobility in patients with Parkinson's disease and other neurological disorders will be significantly more effective and efficient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease
* Ages 50-80
* Currently taking some form of Carbidopa/Levodopa

Exclusion Criteria:

* Significant orthopedic injuries or surgeries
* Deep-Brain-Stimulation surgery
* Any other neurological conditions

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Movement Disorders Clinic at OHSU in Portland Oregon.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
iMOBILITY: the instrumented system for measuring mobility. | 2 years
  Instrumented system for measuring mobility.
  Which measures over a 100 different variables of movement, for example:
  Cadence, Turning Duration, Turning Velocity etc...

CONTACTS AND LOCATIONS:
Overall Officials: Fay Horak, Phd, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Clinical Translational Research Institute, Portland, Oregon, United States